CLINICAL TRIAL: NCT02042391
Title: Risk-stratified Sequential Treatment of Post-transplant Lymphoproliferative Disease (PTLD) With 4 Courses of Rituximab SC Followed by 4 Courses of Rituximab SC, 4 Courses of Rituximab SC Combined With CHOP-21 or 6 Courses of Rituximab SC Combined With Alternating CHOP-21 and DHAOx: The PTLD-2 Trial
Brief Title: Risk-stratified Sequential Treatment of Post-transplant Lymphoproliferative Disease (PTLD) With Rituximab SC and Immunochemotherapy
Acronym: PTLD-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diako Ev. Diakonie-Krankenhaus gemeinnützige GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPTLDSG-IIT-PTLD-2
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Posttransplant Lymphoproliferative Disorder
Keywords: PTLD; CD20-positive; solid organ transplantation
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Oxaliplatin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low-risk (Experimental): All patients will receive rituximab sc on days 1, 8, 15 and 22. Interim staging will be performed around day 50. After interim staging, patients will be considered low-risk if they reached a complete remission with the first 4 applications of rituximab monotherapy or if they reached a partial remission and had a baseline IPI of 0, 1 or 2. Patients considered low-risk will receive rituximab sc consolidation.
  Interventions: Drug: Rituximab sc; Drug: Rituximab sc consolidation
- High risk (Experimental): All patients will receive rituximab sc on days 1, 8, 15 and 22. Interim staging will be performed around day 50. After interim staging, patients will be considered high-risk, if the reached a partial remission and were IPI 3, 4 or 5 at time of diagnosis of PTLD, if they show stable disease or if they had progressive disease but are not recipients of heart or lung transplants. Patients considered high-risk will receive four more applications of rituximab sc combined with CHOP chemotherapy every 3 weeks at days 50, 71, 92 and 113.
  Interventions: Drug: Rituximab sc; Drug: Rituximab sc combined with CHOP chemotherapy
- Very high-risk (Experimental): All patients will receive rituximab sc on days 1, 8, 15 and 22. Interim staging will be performed around day 50. After interim staging, heart and lung transplant recipients and patients with a combination of organs transplanted including a heart or lung transplant who show disease progression during rituximab monotherapy or at interim staging will be considered very high-risk. Patients considered very high-risk will receive six more applications of rituximab sc combined with alternating chemotherapy with CHOP and DHAOx.
  Interventions: Drug: Rituximab sc; Drug: Rituximab sc combined with alternating chemotherapy with CHOP and DHAOx

INTERVENTIONS:
Drug: Rituximab sc — All patients will receive 4 courses of rituximab on days 1, 8, 15 and 22. Rituximab will be administered as a single therapeutic agent at a standard dosage of 375 mg/m2 infused intravenously at day 1. Three subsequent single therapeutic agent applications of rituximab will be administered subcutaneously at a fixed dose of 1400 mg once a week for 3 weeks at days 8, 15 and 22.
  Other Names: Mabthera sc
Drug: Rituximab sc consolidation — Patients considered low-risk will receive four more single therapeutic agent applications of rituximab administered subcutaneously at a fixed dose of 1400 mg once every three weeks at days 50, 71, 92 and 113.
  Other Names: Rituximab sc; Mabthera sc
  Arms: Low-risk
Drug: Rituximab sc combined with CHOP chemotherapy — Patients considered high-risk will receive four more applications of rituximab administered subcutaneously at a fixed dose of 1400 mg combined with CHOP chemotherapy every 3 weeks at days 50, 71, 92 and 113. CHOP chemotherapy will be administered at standard doses: cyclophosphamide 750 mg/m2, adriamycine 50 mg/m2, vincristine 1.4mg/m2 (maximum total dose: 2mg) and prednisone 100mg (at day 1 to 5 of each cycle). Cyclophosphamid, adriamycine and vincristine will be infused intravenously. Prednison will be administered orally in a single dose. At day 3-4 of each treatment cycle either a single dose of 6 mg Peg-GCSF or repetitive doses of 5 µg/kg GCSF until recovery of WBC will be applied subcutaneously, as per institutional practice.
  Other Names: Mabthera sc; Cyclophosphamide; Adriamycine; Vincristin; Prednisone
  Arms: High risk
Drug: Rituximab sc combined with alternating chemotherapy with CHOP and DHAOx — Patients considered very high-risk will receive six more applications of rituximab sc at a fixed dose of 1400 mg combined with chemotherapy every 3 weeks. Chemotherapy is CHOP at days 50, 92 and 134 (cyclophosphamide IV 750 mg/m2, adriamycine IV 50 mg/m2, vincristine IV 1.4mg/m2 (maximum total dose: 2mg) and prednisone PO 100mg (at day 1 to 5 of each cycles). Chemotherapy is DHAOx at days 71, 113 and 155 (oxaliplatin (130 mg/m2, day 1) and cytarabine (ARA-C, 2x 1000 mg/m2 at day 2) dexamethasone PO (40 mg/m2, day 1)), as per institutional practice. At day 3-4 of each treatment cycle either a single dose of 6 mg Peg-GCSF or repetitive doses of 5 µg/kg GCSF until recovery of WBC will be applied subcutaneously, as per institutional practice.
  Other Names: Mabthera sc; Cyclophosphamide; Adriamycine; Vincristin; Prednisone; Oxaliplatin; Cytarabine; Ara-C; Dexamthasone
  Arms: Very high-risk

SUMMARY:
Post-transplant lymphoproliferative disorders (PTLD) differ clinically from lymphoma in the general (immunocompetent) population due to their higher incidence and their frequent association with Epstein-Barr virus. Previous clinical trials have shown their remarkably good response to rituximab as well as to chemotherapy.

The PTLD-1 trial demonstrated the efficacy and safety of sequential immunochemotherapy with 4 courses of rituximab IV followed by 4 cycles of CHOP chemotherapy. Compared to trials of rituximab monotherapy in PTLD, median overall survival was extended from 2.4 to 6.5 years. Compared to previous trials of chemotherapy, complications were reduced. In addition, we noted that those patients who already had a good response to the first four cycles of rituximab did better overall than those who did not. As a consequence, the PTLD-1/3 trial introduced risk-stratification in sequential treatment according to the response to the first 4 courses of rituximab monotherapy. Those patients with a complete remission went on to receive four further courses of rituximab whereas those who did not received rituximab and CHOP chemotherapy. Interim results have demonstrated that it is safe to restrict chemotherapy treatment in this manner and thus established the concept of treatment stratification based on the response to rituximab.

The PTLD-2 trial is the next step in the development of this strategy. Compared to the PTLD-1/3 trial, the key difference is the use of subcutaneous instead of intravenous rituximab application. Interim results from an ongoing trial of patients with follicular lymphoma (NCT01200758) have shown that subcutaneous administration results in increased blood levels and in non-inferior remission rates. Furthermore, the stratification strategy is refined based on observations from the previous PTLD-1 and PTLD1/3 trials: Risk groups are now defined not only based on response to rituximab therapy but also on the international prognostic index (IPI, a well-established lymphoma risk score) and the transplanted organ. The major advantage of this new stratification is an extended low-risk group that is eligible for subcutaneous rituximab monotherapy: Patients with a low risk of disease progression, defined as those who achieve a complete remission after the first four courses of subcutaneous rituximab monotherapy and those with an IPI of 0 to 2 who achieve a partial remission at interim staging, will go on with rituximab monotherapy. Patients with high IPI who achieve a partial remission, patients with stable disease at interim staging and non-thoracic transplant recipients with progressive disease at interim staging will be considered high risk. These patients will go on with 4 cycles of rituximab plus CHOP chemotherapy similar to the PTLD-1/3 protocol. Thoracic transplant recipients refractory to rituximab will be considered very high risk and will go on with rituximab subcutaneous plus alternating chemotherapy with CHOP and DHAOx.

The trial hypothesis is that the new protocol will improve the event-free survival, a measure integrating unfavorable events such as death, disease progression and treatment complications, particularly infections, in the low risk-group compared to the results of the PTLD-1 trial. In very high-risk patients data from the PTLD-1 and PTLD-1/3 trial have shown that the current treatment is not sufficient to control the disease. Death due to disease progression was observed in more than 80% of patients. Here, rituximab combined with alternating chemotherapy cycles of CHOP and DHAOx (+GCSF) may increase treatment efficacy with an acceptable toxicity profile.

In summary, the PTLD-2 trials tests if the substitution of subcutaneous for intravenous rituximab and an updated stratification strategy that deescalates treatment for those at low risk and escalates treatment for those at very high risk can further improve the overall efficacy and safety of PTLD therapy.

ELIGIBILITY:
Inclusion Criteria:

* CD20-positive PTLD with or without EBV association, confirmed after biopsy or resection of tumor
* Measurable disease of > 2 cm in diameter and/or bone marrow involvement
* Patients having undergone heart, lung, liver, kidney, pancreas, small intestine transplantation or a combination of the organ transplantations mentioned
* ECOG ≤ 2
* Clinically insufficient response to an upfront reduction of immunosuppression with or without antiviral therapy
* Age at least 18 years
* Not legally incapacitated
* Written informed consent from the trial subject has been obtained

Exclusion Criteria:

* Complete surgical extirpation of the tumor or irradiation of residual tumor masses
* Upfront treatment with rituximab or chemotherapy
* Known allergic reactions against foreign proteins
* Concomitant diseases, which exclude the administration of therapy as outlined by the study protocol
* Meningeal and CNS involvement
* Known to be HIV-positive
* Pregnant women and nursing mothers
* Failure to use highly-effective contraceptive methods
* Persons held in an institution by legal or official order
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Life expectancy less than 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Event free survival (EFS) of low-risk patients in the intention to treat population with following definitions for low-risk and event: | two years
  Time from start of treatment to event with following definitions for low-risk and event:
  1. Low-risk:
     * all patients in complete remission at interim staging, i.e. 4 weeks after the four weekly courses of rituximab SC monotherapy
     * all patients in partial remission at interim staging with an initial international prognostic index (IPI) of 0,1 or 2
  2. Events:
     * any grade III or IV infection during the treatment period
     * treatment discontinuation from any reason
     * disease progression at any time
     * death from any reason

SECONDARY OUTCOMES:
Overall survival | Two years
Time to progression | two years
Progression-free survival | two years
Response at interim staging | day 50
Response after full treatment | three months
Duration of response | two years
Treatment-related mortality | three months

OTHER OUTCOMES:
Frequency of grade III and IV leucocytopenia and grade III and IV infections by treatment group | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Ralf U Trappe, Dr. med.-, Principal Investigator — DIAKO Bremen
Locations (18):
- Germany (18):
  - Uniklinik RWTH Aaachen Klinik für Onkologie, Hämatologie und Stammzell-transplantation Med. Klinik IV, Aachen
  - Charite Universitätsmedizin Berlin Campus Mitte, Medizinische Klinik mit Schwerpunkt Hämatologie und Onkologie, Berlin
  - Charité - Universitätsmedizin Berlin CCM Medizinische Klinik m. S. Nephrologie, Berlin
  - Universitätsklinikum Bonn Med. Klinik III/ZIM Hämatologie/Onkologie, Bonn
  - DIAKO Bremen gGmbH, Klinik für Hämatologie und Onkologie, Bremen
  - Universitätsklinikum Erlangen Med. Klinik 5 Hämatologie und Intern. Onkologie, Erlangen
  - Universitätsklinikum Essen Klinik für Hämatologie, Essen
  - Malteser Krankenhaus St. Franziskus-Hospital Med. Klinik 1, Flensburg
  - Universitätsklinikum Frankfurt Med. Klinik III, Nephrologie, Frankfurt am Main
  - Universitätsklinikum Gießen Med. Klinik IV, Giessen
  - Medizinische Hochschule Hannover Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation, Hanover
  - II. Medizinische Klinik, Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsmedizin der Johannes-Gutenberg-Universität III. Medizinische Klinik, Mainz
  - Klinikum der Universität München-Großhadern Med. Klinik III, München
  - Klinikum Oldenburg gGmbH Klinik für Innere Medizin II, Oldenburg
  - Klinikum Passau II. Med. Klinik, Passau
  - Universitätsmedizin Rostock Klinik für Innere Medizin III Hämatologie, Onkologie, Palliativmedizin, Rostock
  - Klinikum Stuttgart Klinik für Hämatologie und int. Onkologie, Stuttgart

REFERENCES:
- [Background] Trappe R, Oertel S, Leblond V, Mollee P, Sender M, Reinke P, Neuhaus R, Lehmkuhl H, Horst HA, Salles G, Morschhauser F, Jaccard A, Lamy T, Leithauser M, Zimmermann H, Anagnostopoulos I, Raphael M, Riess H, Choquet S; German PTLD Study Group; European PTLD Network. Sequential treatment with rituximab followed by CHOP chemotherapy in adult B-cell post-transplant lymphoproliferative disorder (PTLD): the prospective international multicentre phase 2 PTLD-1 trial. Lancet Oncol. 2012 Feb;13(2):196-206. doi: 10.1016/S1470-2045(11)70300-X. Epub 2011 Dec 13. PMID 22173060
- [Background] Choquet S, Oertel S, LeBlond V, Riess H, Varoqueaux N, Dorken B, Trappe R. Rituximab in the management of post-transplantation lymphoproliferative disorder after solid organ transplantation: proceed with caution. Ann Hematol. 2007 Aug;86(8):599-607. doi: 10.1007/s00277-007-0298-2. Epub 2007 May 24. PMID 17522862
- [Background] Choquet S, Trappe R, Leblond V, Jager U, Davi F, Oertel S. CHOP-21 for the treatment of post-transplant lymphoproliferative disorders (PTLD) following solid organ transplantation. Haematologica. 2007 Feb;92(2):273-4. doi: 10.3324/haematol.10595. PMID 17296588
- [Background] Oertel SH, Verschuuren E, Reinke P, Zeidler K, Papp-Vary M, Babel N, Trappe RU, Jonas S, Hummel M, Anagnostopoulos I, Dorken B, Riess HB. Effect of anti-CD 20 antibody rituximab in patients with post-transplant lymphoproliferative disorder (PTLD). Am J Transplant. 2005 Dec;5(12):2901-6. doi: 10.1111/j.1600-6143.2005.01098.x. PMID 16303003
- [Result] Zimmermann H, Koenecke C, Dreyling MH, Pott C, Duhrsen U, Hahn D, Meidenbauer N, Hauser IA, Rummel MJ, Wolf D, Heuser M, Schmidt C, Schlattmann P, Ritgen M, Siebert R, Oschlies I, Anagnostopoulos I, Trappe RU. Modified risk-stratified sequential treatment (subcutaneous rituximab with or without chemotherapy) in B-cell Post-transplant lymphoproliferative disorder (PTLD) after Solid organ transplantation (SOT): the prospective multicentre phase II PTLD-2 trial. Leukemia. 2022 Oct;36(10):2468-2478. doi: 10.1038/s41375-022-01667-1. Epub 2022 Aug 16. PMID 35974101
- See also: PTLD-2 trial full text article including supplements (open access) — https://rdcu.be/cT7Qu